CLINICAL TRIAL: NCT02967250
Title: 7T Magnetic Resonance Spectroscopy Monitoring Brain Bioenergetics in Parkinson's Disease and Response to Repeated Oral UDCA Treatment
Brief Title: Brain Bioenergetics in Parkinson's Disease and Response to Repeated Oral UDCA Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEUR-2016-18222
Record Dates: First submitted 2016-09-13; First posted 2016-11-18 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ursodeoxycholic acid treatment (Experimental): Each subject will receive UDCA intervention for six weeks.
  Interventions: Drug: ursodeoxycholic acid

INTERVENTIONS:
Drug: ursodeoxycholic acid — Subjects will be provided ~50mg/kg/day (based on the use of 250 and 500mg capsules) of UDCA to be divided into 3 equal daily doses and titrated up over ~2 weeks to a stable dose for 4 weeks.
  Other Names: Ursodiol

SUMMARY:
The objective of this study is to understand the bioenergetic impairments that underlie Parkinson's disease (PD) and evaluating treatments that may improve abnormal mitochondrial function that is present in PD. The hypothesis is that repeated oral dosing of UDCA will result in increased brain ATP levels in individuals with Parkinson's disease (PD). The specific aims are 1.) to measure plasma UDCA levels in individuals with PD at baseline and after four weeks of repeated high doses of oral UDCA (50mg/kg/day) and 2.) to measure cortical bioenergetic profile and ATPase activity (as ascertained through MRS) in those with PD at baseline and at four weeks after repeated high doses of oral UDCA (50mg/kg/day) simultaneously. Secondary aims are to characterize oral UDCA pharmacokinetics and develop a pharmacokinetic/pharmacodynamic model to characterize the relationship between peripheral measurements of UDCA (and associated conjugates) and peripheral measures and/or central (brain) bioenergetic measurements.

DETAILED DESCRIPTION:
The objective of this study is to understand the bioenergetic impairments that underlie Parkinson's disease (PD) and evaluating treatments that may improve abnormal mitochondrial function that is present in PD. High field - 7 tesla (T) - magnetic resonance spectroscopy (MRS) is able to non-invasively assess for changes in brain energetics and will be used to evaluate the effects that repeated oral doses of the mitochondrial enhancer ursodeoxycholic acid (UDCA) has on brain bioenergetics derived from MRS measurements. This study will combine results obtained using MRS brain scans along with peripheral measurements of bile acids (e.g., total UDCA). This research will require at least 2 visits: baseline evaluation and at approximately 6 weeks after subjects are on a stable oral dose for 4 weeks. Participants will provide their medical history during the first visit, and undergo a physical examination and rating scale each visit (duration: ~1 hour) as well as a brain MRI scan (1-1.5 hours). Blood will be obtained at both visits to monitor for adverse effects as well as to assess for changes in bile acids from orally administered UDCA. If additional funding is obtained we may have another visit added between the first and second assessments to obtain additional blood measurements and MRS data.

Since there is extensive animal and cell model data supporting the rationale for a therapeutic trial of UDCA in PD, and because MRS methods can non-invasively detect changes in brain chemistry we propose a study to evaluate the effects of a 4-6 weeks of high-dose oral UDCA on central (brain) and peripheral measures (through MRS and blood measurements, respectively) in individuals with PD and healthy controls. The hypothesis and specific aims are as follows:

Hypothesis: Repeated oral dosing of UDCA will result in increased brain ATP levels in individuals with Parkinson's disease (PD).

Specific Aims:

1. Measure plasma UDCA levels in individuals with PD at baseline and after four weeks of repeated high doses of oral UDCA (50mg/kg/day).
2. Measure cortical bioenergetic profile and ATPase activity (as ascertained through MRS) in those with PD at baseline and at four weeks after repeated high doses of oral UDCA (50mg/kg/day) simultaneously with Aim 1.

Secondary Aims:

1. Characterize oral UDCA pharmacokinetics
2. Develop a pharmacokinetic/pharmacodynamic model to characterize the relationship between peripheral measurements of UDCA (and associated conjugates) and peripheral measures and/or central (brain) bioenergetic measurements.

ELIGIBILITY:
Inclusion Criteria:

1. All participants must be 18 years or older.
2. All enrollees must understand and cooperate with requirements of the study and be able to provide written informed consent
3. Individuals with medically stable mild to moderate Parkinson's disease or healthy controls (as determined by enrolling investigator)
4. All participants must not have taken UDCA for 4 weeks prior to the study.
5. Absence of dementia in all subjects, as determined by pre-scanning cognitive assessment.

Exclusion Criteria:

1. Inability to undergo MRI scanning without sedation and other MRI counterindications, such as metal in the body.
2. Medically unstable conditions
3. Pregnant or lactating or those women of child-bearing age that are not using acceptable forms of contraception
4. Unable to adhere to study protocol as determined by the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change in ATP concentration | prior to intervention and at 6 weeks of intervention
  measurement of ATP concentrations in brain using 7T MRS

SECONDARY OUTCOMES:
UDCA pharmacokinetics | at 6 weeks of intervention
  measurement of UDCA concentration in plasma will be used to determine pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Coles, PhD, Principal Investigator — University of Minnesota; Paul Tuite, MD, Principal Investigator — University of Minnesota
Locations (1):
- Center for Magnetic Resonance Research, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided